CLINICAL TRIAL: NCT05347251
Title: Effects of Cervicothoracic Mobility Program on Pain, Range of Motion and Function in Patients With Chronic Back Pain
Brief Title: Effects of Cervicothoracic Mobility Program on Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/22/0137 Amna
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Back Pain
Keywords: Back pain; Cervical mobilization; Thoracic mobilization
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Cervicothoracic mobility program
  Interventions: Other: Cervicothoracic mobility program
- Group B (Other): Conventional Treatment
  Interventions: Other: Conventional Treatment

INTERVENTIONS:
Other: Cervicothoracic mobility program — Participants in this group will receive mobilization at a cervical and thoracic level along with conventional physical therapy protocol like Hot packs and exercise therapy.
  At the cervical, PA glides (central) and transverse glides will be given for mobilization.
  At thoracic, PA glides (central) and transverse glides will be given for mobilization.
  Exercise therapy includes stretching and strengthening both cervical and thoracic muscles. At the cervical level, neck isometric (flexion, extension, side bending) will be given to patients to enhance strengthening, and neck
  stretching exercises (flexors, extensors, side benders
  and rotators) will perform as well. Similarly, at the thoracic
  level, strengthening and stretching of thoracic muscle will be performed
  Arms: Group A
Other: Conventional Treatment — It will be the control group. The participants who will be allocated in this group receive the only conventional physical therapy protocol (Hot pack and exercise therapy). Exercise therapy includes stretching and strengthening of neck and upper back muscles. At the cervical level, neck isometric (flexion, extension, side bending) will be given to patients to enhance strengthening, and neck stretching exercises (flexors,
  extensors, side benders, and rotators) will perform
  as well. Similarly at the thoracic level, strengthening and stretching of thoracic muscle will be performed.
  Arms: Group B

SUMMARY:
The study will be a randomized control trial to determine the effects of the cervicothoracic mobility program on pain, range of motion, and function in patients with chronic back pain. The purposive sampling technique will be used. A sample of 44 patients will be taken and divided into two groups each with 22 patients. Group A will be the experimental group and group B will be the control group. The experimental group will receive cervical mobility and thoracic mobility along with conventional physical therapy protocols like hot packs and exercise therapy protocol. Group B will be the control group and will receive the conventional physical therapy protocol like the hot pack and exercise therapy protocol. Exercise therapy includes the strengthening and stretching exercises of both neck and back muscles.

The session will be around 40 to 45 min for each patient with three sessions per week on alternate days. A total of 3-week treatment program will be given to the patients and an assessment of the patient's pain, range of motion, and function with NPRS (numeric pain rating scale), goniometer, and ODI (Oswestry disability index) will be done at the baseline and after the completion of treatment at three weeks.

DETAILED DESCRIPTION:
Chronic back pain is usually age-related, but can also result from a prior injury. The most common causes include arthritis of the spine, a sedentary lifestyle, and any injury or disc-related problems. Joint mobilization is a physical therapy technique designed to relieve pain and muscle spasms, release tension and improve flexibility in a joint. The aim of this study is to determine the effects of the cervicothoracic mobility program on pain, range of motion, and function in patients with chronic back pain. The study will be a randomized control trial to determine the effects of the cervicothoracic mobility program on pain, range of motion and function in patients with chronic back pain. The purposive sampling technique will be used. A sample of 44 patients will be taken and divided into two groups each with 22 patients. Group A will be the experimental group and group B will be the control group. The experimental group will receive cervical mobility and thoracic mobility along with conventional physical therapy protocols like a hot pack and exercise therapy protocol. Group B will be the control group and will receive the conventional physical therapy protocol like hot pack and exercise therapy protocol. Exercise therapy includes the strengthening and stretching exercises of both neck and back muscles. The session will be around of 40 to 45 min on each patient with three sessions per week on alternate days. A total of 3-week treatment program will be given to the patients and an assessment of the patient's pain, range of motion and function with NPRS (numeric pain rating scale), goniometer and ODI (Oswestry disability index) will be done at the baseline and after the completion of treatment at three weeks.

ELIGIBILITY:
Inclusion Criteria:

* Both genders.
* Age 18-50 years. NPRS between 3 and 6
* Subjects diagnosed with chronic back pain with minimum 6 months of chronicity
* ODI score 21 to 40
* There should be no radiating pain to legs of participants.

Exclusion Criteria:

* Patients with Systemic soft tissue disease and bony disease will be excluded from the study.
* Pregnant women will be excluded from the study.
* Patients with previous orthopedic and neurosurgical surgery will be excluded from the study.
* Patients with any Red flags (Ankylosing spondylitis, spondylolisthesis, Slipped discs, spinal tumor, spinal stenosis, cauda equine syndrome, and spine infection) will be excluded.
* Patients with a positive Faber test for SIJ dysfunction will be excluded

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
NPRS | 3rd Week
  Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. Where 0 indicate no pain and 10 indicate severe pain
ODI | 3rd Week
  The Oswestry Disability Index is an extremely important tool that researchers and disability evaluators use tomeasure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools
Goniometer | 3rd Week
  A goniometer is an instrument which measures the available range of motion at a joint.
  (Also mention all information which ROM u want to check)

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil Ur Rehman, PhD, Principal Investigator — Riphah International University
Locations (1):
- Physiotherapy department of Syed medical complex Sialkot, Sialkot, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Husky MM, Ferdous Farin F, Compagnone P, Fermanian C, Kovess-Masfety V. Chronic back pain and its association with quality of life in a large French population survey. Health Qual Life Outcomes. 2018 Sep 26;16(1):195. doi: 10.1186/s12955-018-1018-4. PMID 30257670
- [Background] Ganesan S, Acharya AS, Chauhan R, Acharya S. Prevalence and Risk Factors for Low Back Pain in 1,355 Young Adults: A Cross-Sectional Study. Asian Spine J. 2017 Aug;11(4):610-617. doi: 10.4184/asj.2017.11.4.610. Epub 2017 Aug 7. PMID 28874980
- [Background] Sung YB, Lee JH, Park YH. Effects of thoracic mobilization and manipulation on function and mental state in chronic lower back pain. J Phys Ther Sci. 2014 Nov;26(11):1711-4. doi: 10.1589/jpts.26.1711. Epub 2014 Nov 13. PMID 25435683
- [Background] Rubinstein SM, de Zoete A, van Middelkoop M, Assendelft WJJ, de Boer MR, van Tulder MW. Benefits and harms of spinal manipulative therapy for the treatment of chronic low back pain: systematic review and meta-analysis of randomised controlled trials. BMJ. 2019 Mar 13;364:l689. doi: 10.1136/bmj.l689. PMID 30867144
- [Background] Khan S, Al Torairi N, Shamsi S. Comparative Study Of Snags And Maitland's Mobilization In Chronic Low Back Pain. European Journal of Physical Education and Sport Science. 2018.
- [Background] Sahin N, Karahan AY, Albayrak I. Effectiveness of physical therapy and exercise on pain and functional status in patients with chronic low back pain: a randomized-controlled trial. Turk J Phys Med Rehabil. 2017 Aug 9;64(1):52-58. doi: 10.5606/tftrd.2018.1238. eCollection 2018 Mar. PMID 31453489
- [Background] Divya, Parveen A, Nuhmani S, Ejaz Hussain M, Hussain Khan M. Effect of lumbar stabilization exercises and thoracic mobilization with strengthening exercises on pain level, thoracic kyphosis, and functional disability in chronic low back pain. J Complement Integr Med. 2020 Jul 27;18(2):419-424. doi: 10.1515/jcim-2019-0327. PMID 32712591
- [Background] Thomas JS, Clark BC, Russ DW, France CR, Ploutz-Snyder R, Corcos DM; RELIEF Study Investigators. Effect of Spinal Manipulative and Mobilization Therapies in Young Adults With Mild to Moderate Chronic Low Back Pain: A Randomized Clinical Trial. JAMA Netw Open. 2020 Aug 3;3(8):e2012589. doi: 10.1001/jamanetworkopen.2020.12589. PMID 32756930
- [Background] Lim C-G. Comparison of the effects of joint mobilization, gym ball exercises, and breathing exercises on breathing pattern disorders and joint position sense in persons with chronic low back pain. Physical Therapy Rehabilitation Science. 2020;9(1):25-35.
- [Background] Herman PM, Whitley MD, Ryan GW, Hurwitz EL, Coulter ID. The impact of patient preferences and costs on the appropriateness of spinal manipulation and mobilization for chronic low back pain and chronic neck pain. BMC Musculoskelet Disord. 2019 Nov 7;20(1):519. doi: 10.1186/s12891-019-2904-6. PMID 31699077
- [Background] Yang D, Park S, Kang J, Kim J, Jung D, Kim Y, et al. The effect of spine mobilization technique on balance and the low back pain disability index of patients with chronic back pain. Journal of The Korean Society of Integrative Medicine. 2018;6(4):139-48
- [Derived] Naseer A, Ur Rehman SS, Fatima G, Ikram M. Effects of cervicothoracic mobility programme on pain, range of motion and function in patients with chronic back pain. J Pak Med Assoc. 2024 Jul;74(7):1291-1295. doi: 10.47391/JPMA.10939. PMID 39028057